CLINICAL TRIAL: NCT05561010
Title: Is There a Difference in the Analgesic Response to Intra-articular Bupivacaine Injection in People With Knee Osteoarthritis Pain With or Without Central Sensitisation?: a Feasibility Randomised Controlled Trial
Brief Title: Understanding Pain Mechanisms in Knee Osteoarthritis
Acronym: UP-KNEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); Versus Arthritis (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19OR016
Record Dates: First submitted 2020-12-15; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee; Chronic Pain
Keywords: Knee osteoarthritis; Chronic pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular injection of bupivacaine (Experimental): 5 ml of bupivacaine (0.25% w/v)
  Interventions: Drug: Intra-articular injection of bupivacaine in the knee joint
- Intra-articular injection of sodium chloride (Placebo Comparator): 5 ml of sodium chloride (9mg/ml, 0.9% solution for injection)
  Interventions: Drug: Intra-articular injection of placebo in the knee joint

INTERVENTIONS:
Drug: Intra-articular injection of bupivacaine in the knee joint — 25 participants will be allocated to the bupivacaine arm.
  Other Names: Bupivacaine hydrochloride
  Arms: Intra-articular injection of bupivacaine
Drug: Intra-articular injection of placebo in the knee joint — 25 participants will be allocated to the placebo arm.
  Other Names: Sodium chloride
  Arms: Intra-articular injection of sodium chloride

SUMMARY:
UP-KNEE study is a feasibility, double-blind, placebo-controlled randomised parallel study in participants with radiographically defined knee OA, and with self-reported chronic knee pain.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee joint is a common cause of chronic pain, disability and impaired quality of life. Knee OA affects ~ 1 in 5 adults over 45 years, with many requiring major knee surgery to alleviate pain and restore mobility. However, > 1 in 5 patients will continue to suffer from pain despite surgery. It remains largely unknown who will fail to respond, and why.

Chronic postoperative pain may be linked to a particular type of pain, that is not only driven by the joint damage itself but by changes in the central nervous system (central pain). Several lines of evidence support this idea, but there is a need for a better understanding of the underlying mechanisms as well as a better tool to differentiate between peripherally- and centrally-augmented knee pain in order to identify who will benefit the most from knee surgery.

To this end, the proposed research is a feasibility study aiming to provide proof of concept for a future main trial. The study combines the diagnostic power of non-invasive imaging with experimental approaches to investigate central pain by modelling the peripheral effects of knee surgery. This will provide novel insights into the contribution of peripheral and central pain mechanisms in knee OA which can pave the way for better treatment results.

This study is expected to last for one year. It is funded by Versus Arthritis Pain Centre and forms part of a wider scientific project aiming at increasing knowledge and understanding of OA pain.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically defined OA knee changes (K/L > 2);
* Must have self-reported knee pain (measuring at least 30 mm to 80 mm on a 100 mm VAS for rest, use or night pain);
* Able to give informed consent;
* Aged 45 years and older;
* All genders;
* Able to perform the six-minute walk test.

Exclusion Criteria:

* Aged less than 45 years;
* Breastfeeding or pregnancy;
* Not having the capacity to consent;
* Non-English speakers;
* Major medical, neurological and psychiatric co-morbidities;
* Hip OA (ipsilateral or contralateral);
* Fibromyalgia;
* Sensory dysfunctional illness;
* Chronic pain conditions other than OA;
* Presence of local or systemic infection or suspicion of infection in the knee joint, overlying soft tissue or elsewhere;
* History of septic arthritis in the knee to be injected;
* Acute haemarthrosis in the joint to be injected;
* Recent trauma within 72 hours;
* Prosthetic joint;
* Presence of broken skin or rash over the area to be injected;
* Severe coagulopathy (can take aspirin or anti-platelets inhibitors such as clopidogrel);
* Any anti-coagulant therapy (e.g. warfarin);
* Severe liver disease or severe kidney disease;
* Known hypersensitivity, allergy or intolerance to local anaesthetic / bupivacaine;
* Recently taken other medicines containing local anaesthetic / bupivacaine within 1 month;
* Surgery planned within 3 months of entry to study;
* Neuropathic pain medications such as opioid analgesics, antiepileptic drugs such as pregabalin / gabapentin, and tricyclic antidepressants such as amitriptyline when taken for neuropathic pain treatment;
* Current or recent intake centrally-active medication (e.g. have recently taken monoamine oxidase inhibitor (MAOI));
* Complete heart block;
* The presence of any contraindication for MRI.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in pain score during the six-minute walk test | From baseline to approximately one hour after intra-articular injection with bupivacaine or placebo
  The change from baseline in pain score using the Visual Analogue Scale during the six-minute walk test.
  (visual analogue scale ranges from 0-100; 0 meaning no pain and 100 worst imaginable pain)
The change from baseline in pain score at rest | From baseline to approximately one hour after intra-articular injection with bupivacaine or placebo
  The change from baseline in pain score using the Visual Analogue Scale at rest. (visual analogue scale ranges from 0-100; 0 meaning no pain and 100 worst imaginable pain)

SECONDARY OUTCOMES:
Quantitative sensory testing (QST) | Baseline and within 30 minutes after intra-articular injection with bupivacaine or placebo
  Correlations between change of pain score and QST findings will be assessed.
Brain functional magnetic resonance imaging (fMRI) | Baseline and 1 hour after intra-articular injection with bupivacaine or placebo
  Correlations between the change of pain score and brain network activity using predefined seeds in the pain processing regions will be assessed.
Magnetic Resonance Imaging Knee Osteoarthritis Score (MOAKS) | Baseline
  Correlations between the change of pain score and the level of joint damage quantified by MOAKS will be assessed. Higher MOAKS indicate worse outcome.
The number of eligible participants who are recruited and randomised to the study | Through study completion, an average of 6 months
  To assess the feasibility of recruitment, the number of eligible participants who are recruited and randomised to the study will be measured.
A study-specific checklist to assess the feasibility of the randomisation process | Through study completion, an average of 6 months
  Evaluation of effective randomisation of participants to the study arms using a study-specific checklist and assessment of the randomisation protocol throughout the study.
A study-specific questionnaire to assess the acceptability of the trial methods | Assessed immediately after the final intervention
  A study-specific questionnaire will be administered to participants to assess the acceptability of the study design and research process.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Brigitte Scammell, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745-1759. doi: 10.1016/S0140-6736(19)30417-9. PMID 31034380
- [Background] Creamer P, Hunt M, Dieppe P. Pain mechanisms in osteoarthritis of the knee: effect of intraarticular anesthetic. J Rheumatol. 1996 Jun;23(6):1031-6. PMID 8782136
- [Background] Hassan BS, Doherty SA, Mockett S, Doherty M. Effect of pain reduction on postural sway, proprioception, and quadriceps strength in subjects with knee osteoarthritis. Ann Rheum Dis. 2002 May;61(5):422-8. doi: 10.1136/ard.61.5.422. PMID 11959766
- [Background] Arendt-Nielsen L, Egsgaard LL, Petersen KK, Eskehave TN, Graven-Nielsen T, Hoeck HC, Simonsen O. A mechanism-based pain sensitivity index to characterize knee osteoarthritis patients with different disease stages and pain levels. Eur J Pain. 2015 Nov;19(10):1406-17. doi: 10.1002/ejp.651. Epub 2014 Dec 29. PMID 25545011
- [Background] Bird SB, Dickson EW. Clinically significant changes in pain along the visual analog scale. Ann Emerg Med. 2001 Dec;38(6):639-43. doi: 10.1067/mem.2001.118012. PMID 11719742
- [Background] Suokas AK, Walsh DA, McWilliams DF, Condon L, Moreton B, Wylde V, Arendt-Nielsen L, Zhang W. Quantitative sensory testing in painful osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2012 Oct;20(10):1075-85. doi: 10.1016/j.joca.2012.06.009. Epub 2012 Jul 13. PMID 22796624
- [Background] Kurien T, Arendt-Nielsen L, Petersen KK, Graven-Nielsen T, Scammell BE. Preoperative Neuropathic Pain-like Symptoms and Central Pain Mechanisms in Knee Osteoarthritis Predicts Poor Outcome 6 Months After Total Knee Replacement Surgery. J Pain. 2018 Nov;19(11):1329-1341. doi: 10.1016/j.jpain.2018.05.011. Epub 2018 Jun 18. PMID 29920331
- [Derived] Zedan Y, Knaggs R, Cooper D, Kurien T, Walsh DA, Auer DP, Scammell BE. Is there a difference in the analgesic response to intra-articular bupivacaine injection in people with knee osteoarthritis pain with or without central sensitisation? Protocol of a feasibility randomised controlled trial. BMJ Open. 2023 Jul 11;13(7):e072138. doi: 10.1136/bmjopen-2023-072138. PMID 37433734